CLINICAL TRIAL: NCT06938984
Title: Human TECAR on Exercise Preconditioning and Post-exercise Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7.083.912
Record Dates: First submitted 2025-03-31; First posted 2025-04-22 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Exercise Recovery
Keywords: TECAR therapy; Post-exercise recovery; Preconditioning

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Sham-control (Sham Comparator): Fake intervention - massaging the quadriceps with one of the Human TECAR probes with the device turned off for 10 minutes, before or after the eccentric exercise protocol depending on randomization
  Interventions: Device: Sham Comparator
- Capacitive mode before exercise (Experimental): Capacitive mode applied to the quadriceps for 10 minutes, before the eccentric exercise (preconditioning)
  Interventions: Device: Capacitive mode before
- Resistive mode before exercise (Experimental): Resistive mode applied to the quadriceps for 10 minutes, before the eccentric exercise (preconditioning)
  Interventions: Device: Resistive mode before
- Capacitive mode after exercise (recovery) (Experimental): Capacitive mode applied to the quadriceps for 10 minutes, after the eccentric exercise (recovery)
  Interventions: Device: Capacitive mode after
- Resistive mode after exercise (recovery) (Experimental): Resistive mode applied to the quadriceps for 10 minutes, after the eccentric exercise (recovery)
  Interventions: Device: Resistive mode after

INTERVENTIONS:
Device: Sham Comparator — Massaging the quadriceps with one of the Human TECAR probes with the device turned off for 10 minutes
  Arms: Sham-control
Device: Capacitive mode before — Capacitive mode applied to the quadriceps for 10 minutes
  Arms: Capacitive mode before exercise
Device: Resistive mode before — Resistive mode applied to the quadriceps for 10 minutes
  Arms: Resistive mode before exercise
Device: Capacitive mode after — Capacitive mode applied to the quadriceps for 10 minutes
  Arms: Capacitive mode after exercise (recovery)
Device: Resistive mode after — Resistive mode applied to the quadriceps for 10 minutes
  Arms: Resistive mode after exercise (recovery)

SUMMARY:
TECAR therapy (Transfer of Energy Capacitive and Resistive) is a type of diathermy that uses radiant energy to generate endogenous heat. However, to the date there are no studies investigating the effects of TECAR therapy on exercise preconditioning and post-exercise recovery in humans. Therefore, the aim of this project is to assess the effects of different treatment protocols of TECAR therapy on. exercise preconditioning and post-exercise recovery in humans

DETAILED DESCRIPTION:
Fifty male healthy volunteers will be enrolled in a randomized, double-blind (participants and assessors), controlled trial. Volunteers will be allocated in 5 groups of 10 participants each: 1 - Sham-control (fake intervention - massaging with one of the Human TECAR probes with the device turned off before or after the eccentric exercise protocol depending on randomization); 2 - Capacitive mode before exercise (preconditioning); 3 - Resistive mode before exercise (preconditioning); 4 - Capacitive mode after exercise (recovery); and 5 - Resistive mode after exercise (recovery). The treatment target will be the knee extensors muscles (quadriceps).

A standardized knee extension eccentric exercise protocol performed in the isokinetic dynamometer (Biodex System 4) will be used in order to exercise induce skeletal muscle fatigue and damage.

Volunteers will be treated with Human TECAR in a single treatment session, with 10 minutes length, that will be carried out immediately before or immediately after the exercise protocol according to the randomization.

ELIGIBILITY:
Inclusion Criteria:

* Physically active male participants;
* Do not present a history of musculoskeletal injury in the regions of the hips, knees and calves in the month preceding the study;
* Are not using pharmacological agents;
* Voluntarily commit to participate in all stages of the study.

Exclusion Criteria:

* Present musculoskeletal or joint injuries during data collection;
* Present history of musculoskeletal injury in the regions of the hips, knees and calves in the month preceding the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men
Enrollment: 50 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength | 48 hours after eccentric exercise
  The muscle strength will be measured through isokinetic dynamometry

SECONDARY OUTCOMES:
Change in muscle strength | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  The muscle strength will be measured through isokinetic dynamometry
Change in CK activity | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  The CK activity will be analyzed from the blood samples collected from the participants through biochemical analysis and using specific reagent kits.
Delayed onset muscle soreness - DOMS | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  DOMS will be assessed through the VAS scale
Temperature | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  Thigh temperature will be assessed through Thermography using the WellVu camera.
Muscular oxygen saturation index | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  It will be measured using near-infrared spectroscopy (NIRS)
Muscular blood flow | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  It will be measured analyzing total hemoglobin in muscle tissue using near-infrared spectroscopy (NIRS)
Muscular effort perception | 5 minutes after the treatment, 5 minutes, 1 hour, 24 hours, 72 hours, and 96 hours after the eccentric exercise protocol
  The CR-100 Effort Perception Scale will be used
Participant satisfaction with the treatment | 96 hours after the eccentric exercise protocol
  The Likert scale will be used

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, Ph.D., M.Sc., PT., Principal Investigator — Nove de Julho University
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available six months after the manuscript publication for five years after that.
Access Criteria: All IPD that underlie results in a publication will be available on reasonable request.